CLINICAL TRIAL: NCT04351347
Title: Clinical Study Evaluating the Efficacy of Ivermectin in Larger Doses in COVID-19 Treatment
Brief Title: The Efficacy of Ivermectin in Larger Doses in COVID-19 Treatment
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ivermecin covid
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: COVID
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Experimental): Ivermectin alone in larger doses
  Interventions: Drug: Ivermectin
- Standard treatment (No Intervention): Standard of care treatment

INTERVENTIONS:
Drug: Ivermectin — ivermectin
  Arms: Ivermectin

SUMMARY:
Efficacy of Ivermectin in larger doses in COVID-19 treatment

DETAILED DESCRIPTION:
Clinical Study Evaluating the Efficacy of Ivermectin in higher doses in COVID-19 treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with covid 19

Exclusion Criteria:

* Allergy or side effects to treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improvement or died | 1 month
  The number of patients with improvement or death

CONTACTS AND LOCATIONS:
Overall Officials: sherief Abd-Elsalam, Ass. Prof., Principal Investigator — Tanta University - Faculty of Medicine
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No